CLINICAL TRIAL: NCT00477139
Title: A Pilot Study Evaluating the Immunologic Status of Patients With HER2+ Breast Cancer
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Dr. Ellie Guardino MD/PhD, Stanford University School of Medicine
Other Study IDs: BRSADJ0009; 97811 (Other: Stanford University Alternate IRB Approval Number); BRSADJ0009 (Other: Stanford University)
Record Dates: First submitted 2007-05-18; First posted 2007-05-22 (Estimated); Last update posted 2011-04-13 (Estimated); Status verified 2011-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a pilot study to gather preliminary data on the baseline immunologic status of patients with HER-2(+) breast cancer and to establish an immune monitoring laboratory for future clinical trial.

DETAILED DESCRIPTION:
This is a pilot study to gather preliminary data on the baseline immunologic status of patients with HER-2(+) breast cancer and to establish an immune monitoring laboratory for future clinical trial. We will ask up to 10 patients with HER-2(+) breast cancer in stable condition and in reasonable health to participate in this study. The study will establish an immune monitoring for correlative studies done in patients with HER-2(+) breast cancer. The immunologic tests that will be done are ELISpot, lymphocyte proliferation, intracellular cytokine staining, lymphocyte immunophenotyping, and ELISA.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years of age
* Histologically documented breast cancer (hormone receptor (ER/PR) status may be either positive or negative) with or without metastatic disease.
* HER-2(+) as determined by one of the following measurements. NOTE: HER-2(+) assessment may have been on initial diagnosis and need not be repeated for metastatic lesions

  * Immunohistochemistry (IHC) 3+, or
  * FISH + (HER-2 gene signal to centromere 17 signal >2)
* No transfusion dependent patients and no transfusion within 30 days of leukopheresis
* Documented labs within 7 days of donation consisting of:

  * WBC > 4.0 K/ul & < 11.0 K/ul
  * platelet count > 150,000/mm3
  * hemoglobin > 11.0 g/dl.
  * Hematocrit > 33 %
* Weight > 110 lbs
* No blood donation in last 8 weeks (blood samples taken for standard of care less then 30 cc/week are acceptable)
* Patients must not have active or unresolved infection.
* No cold or flu sympton at time of donation
* No prior myocardial infarction or active cardiac disease (e.g. congestive heart failure, clinically significant cardiac valvular disease or arrhythmia requiring medications, angina pectoris, uncontrolled hypertension, clinically significant pericardial effusion)
* All patients must give signed written informed consent.
* ECOG Performance Score of 0 or 1.
* Women of childbearing potential must have a negative serum or urine pregnancy test

Exclusion Criteria:

* The presence of another active malignancy
* Pregnant, lactating, or nursing
* Patients with prior myocardial infarction or active cardiac disease (e.g. congestive heart failure, clinically significant cardiac valvular disease or arrhythmia requiring medications, angina pectoris, uncontrolled hypertension, clinically significant pericardial effusion)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: individuals with HER-2 positive breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2009-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ellie Guardino MD/PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States